CLINICAL TRIAL: NCT03086135
Title: Clinical Performance of a New Implant System for Bone Conduction Hearing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBAS5539
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2020-01

CONDITIONS: Deafness; Sensoneural Single Sided; Conductive Hearing Loss; Mixed Hearing Loss
MeSH Terms: conditions — Deafness; Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Bone-conduction hearing device (Experimental): The bone-conduction hearing device Osia system allows a direct bone-conduction through an osseointegrated implant. A magnet allows the external Sound Processor to be placed in the correct position over the implanted system including an inner magnet.
  Interventions: Device: Osia System

INTERVENTIONS:
Device: Osia System — An external Sound Processor captures and digitize the sound which is transferred to the internal implant where it is converted to an electrical signal. The electrical signal is further transferred as a vibration through an osseointegrated implant to the mastoid bone and eventually to the cochlea.

SUMMARY:
To study the initial experience with implanting and fitting the new Bone conduction system in patients with conductive, mixed or Single sided Sensorineural deafness.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (18 years or older)
* Subject with conductive or mixed hearing loss in the ear to be implanted. Bone conduction thresholds with pure tone average (PTA4; mean of 0.5, 1, 2 and 4 kHz) of 55 dB HL.

OR Subject with single-sided sensorineural deafness who is a candidate for Baha surgery. Air conduction thresholds with a pure tone average PTA4 of 20 dB HL (mean of 0.5, 1, 2 and 3 kHz) in the good ear OR subject who is indicated for an AC CROS but-for some reason-cannot or will not use an AC CROS (Air Conduction-Contralateral Routing of Signal).

* Signed informed consent
* Previous experience from amplified sound though a non-surgical solution. (For example but not limited to Hearing aid, CROS device, Bone conductional hearing device on headband/ softband)

Exclusion Criteria:

* Uncontrolled diabetes as judged by the investigator.
* Condition that could jeopardise osseointegration and/or wound healing (e.g. osteoporosis, psoriasis, long-term systemic use of corticosteroids) or condition that may have an impact on the outcome of the investigation as judged by the investigator.
* Insufficient bone quality and quantity for implantation of a BI300 Implant.
* Subject that has received radiotherapy in the area of implantation, or is planned for such radiotherapy during the study period
* Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator
* Unable to follow investigational procedures, e.g. to complete quality of life scales.
* Participation in another clinical investigation with pharmaceutical and/or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Mylanus, Prof., Principal Investigator — Radboud Univerity Medical centre; Robert Briggs, Prof., Principal Investigator — The Royal Victorian Eye and Ear Hospita; Susan Arndt, Prof., Principal Investigator — Universitätsklinikum Freiburg; Piotr Skarżyński, Ass.Prof., Principal Investigator — Center of Hearing and Speech; Henry Alexander Arts, Prof., Principal Investigator — University of Michigan
Locations (5):
- University of Michigan, Ann Arbor, Michigan, United States
- The Royal Victorian Eye and Ear Hospital, East Melbourne, Victoria, Australia
- University Medical Center Freiburg, Freiburg im Breisgau, Baden-Wurttemberg, Germany
- Radboud University Medical Center, Nijmegen, Netherlands
- World Hearing Center Institute of Physiology and Pathology of Hearing, Kajetany, Nadarzyn, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bone-conduction Hearing Device
Started | 51
Completed | 48
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 51
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 9
  United States | 10
  Poland | 10
  Australia | 12
  Germany | 10

OUTCOME MEASURES:

1. Primary Outcome: Hearing Performance: Threshold Audiometry, Pure Tone Average of 4 Frequencies, PTA4, Unaided Versus OSIA System at 3 Months
Description: The change of hearing performance from the unaided hearing situation before surgery to the aided hearing situation with the OSIA system at 3 month, measured as free-field hearing test; Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz) is presented. A Pure Tone Average (PTA) refers to the average of hearing threshold levels at a set of specified frequencies: typically 500, 1000, 2000 and 4000 Hz. This value gives a snapshot of an individual's hearing level. If PTA is <25 dB, the overall hearing would be considered to be within normal limits. With a PTA of 95 dB, the hearing would be considered in the profound range. The units reported for PTA4 are decibels (dB). The results presented here are the difference of PTA4 unaided and PTA4 aided with the Osia system. An uaided PTA4 values should be higher than a aided PTA4 if the hearing device is effective. A lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: Baseline before surgery, 3 months after surgery
Measure: Mean (Standard Deviation); unit: dB (Decibel)
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 49
dB (Decibel) | -25.8 (9.1)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; PTA4 at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

2. Primary Outcome: Adaptive Speech Recognition in Noise, Unaided Versus OSIA System at 3 Months.
Description: The change of hearing performance from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 3 months measured as free field hearing test Adaptive speech recognition in noise, is presented. Adaptive speech recognition in noise was measured as Signal to Noise Ratio (SNR). The noise was kept constant at 65 dB SPL and the speech was adapted in dB steps to establish the Speech-to-Noise Ratio (SNR) providing a 50% level of understanding. A ratio of 0 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A negative SNR-value reflects the ability to correctly hear sentences below 65 dB, for example if 50% of the speech is received correctly at 55 dB the SNR value is -10. A positive SNR-value (Speech to Noise Ratio) reflects the ability to correctly hear sentences presented above 65 dB. A lower or more negative score is more desirable and reflects abetter hearing in a noisy enviroment.
Time Frame: Baseline before surgery, 3 months after surgery
Measure: Mean (Standard Deviation); unit: SNR (Speech in Noise Ratio)
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 48
SNR (Speech in Noise Ratio) | -13.3 (8.3)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Speech in noise at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

3. Secondary Outcome: Hearing Performance: Threshold Audiometry, Pure Tone Average, PTA4, Unaided Versus OSIA System at 4 Weeks, 6 and 12 Months
Description: The change of hearing performance from the unaided hearinhg situation before surgery to the aided hearing situation with the OSIA system at 4 weeks, 6 and 12 months, measured as free-field hearing test: Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz) is presented. A Pure Tone Average (PTA) refers to the average of hearing threshold levels at a set of specified frequencies: typically 500, 1000, 2000 and 4000 Hz. This value gives a snapshot of an individual's hearing level. If PTA is <25 dB, the overall hearing would be considered to be within normal limits. With a PTA of 95 dB, the hearing would be considered in the profound range. The units reported for PTA4 are decibels (dB). The results presented here are the difference of PTA4 unaided and PTA4 aided with the Osia system. An uaided PTA4 values should be higher than a aided PTA4 if the hearing device is effective. A lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: Baseline before surgery, 4 weeks, 6 and 12 months after surgery
Population: Some subjects did not perform the test at one or more visits.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
dB
  4 weeks | -24.9 (9.4)
  6 months: number analyzed (Participants) | 49
  6 months | -27.9 (9.1)
  12 months: number analyzed (Participants) | 46
  12 months | -30.4 (8.9)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; PTA4 at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; PTA4 at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; PTA4 at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

4. Secondary Outcome: Hearing Performance: Threshold Audiometry Individual Frequences, Unaided Versus OSIA System at 4 Weeks, 3, 6 and 12 Months
Description: The change of hearing performance from the unaided hearing situation before surgery to the aided hearing situation with the OSIA system at 4 weeks, 3, 6 and 12 months, measured as free-field hearing test: Threshold audiometry (0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz) is presented. This value gives a snapshot of an individual's hearing level. If PTA is <25 dB, the overall hearing would be considered to be within normal limits. With a PTA of 95 dB, the hearing would be considered in the profound range. The units reported for PTA4 are decibels (dB). The results presented here are the difference of the unaided hearing level expressed in dB and the hearing level aided with the Osia system at different time points. An unaided value should be higher than a aided if the hearing device is effective. A lower or more negative score is therefor more desirable and reflects a better ability to hear at the specified frequency.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months after surgery.
Population: 750, 1500 and 8000 Hz were not included in the eCRF for free-field threshold audiometry test due to an error when the first six subjects entered the study. Measurements at these frequencies were therefore not performed at the first visits. In addition; not all subjects performed the test at all frequencies at all visits.
Measure: Mean (Standard Deviation); unit: dB (Decibel)
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
dB (Decibel)
  4 weeks: 250 Hz | -10.3 (12.9)
  4 weeks: 500 Hz | -23.3 (11.1)
  4 weeks: 750 Hz: number analyzed (Participants) | 43
  4 weeks: 750 Hz | -28.3 (12.1)
  4 weeks: 1000 Hz | -26.4 (11.2)
  4 weeks: 1500 Hz: number analyzed (Participants) | 44
  4 weeks: 1500 Hz | -24.2 (12.1)
  4 weeks: 2000 Hz | -23.8 (11.5)
  4 weeks: 3000 Hz | -24.7 (11.3)
  4 weeks: 4000 Hz | -26.1 (10.5)
  4 weeks: 6000 Hz: number analyzed (Participants) | 49
  4 weeks: 6000 Hz | -29.6 (11.3)
  4 weeks: 8000 Hz: number analyzed (Participants) | 38
  4 weeks: 8000 Hz | -29.8 (12.5)
  3 months: 250 Hz: number analyzed (Participants) | 49
  3 months: 250 Hz | -10.8 (13.1)
  3 months: 500 Hz: number analyzed (Participants) | 49
  3 months: 500 Hz | -23.9 (11.3)
  3 months: 750 Hz: number analyzed (Participants) | 43
  3 months: 750 Hz | -28.5 (12.1)
  3 months: 1000 Hz: number analyzed (Participants) | 49
  3 months: 1000 Hz | -27.4 (11.9)
  3 months: 1500 Hz: number analyzed (Participants) | 43
  3 months: 1500 Hz | -25.1 (10.6)
  3 months: 2000 Hz: number analyzed (Participants) | 49
  3 months: 2000 Hz | -24.9 (11.0)
  3 months: 3000 Hz: number analyzed (Participants) | 49
  3 months: 3000 Hz | -26.1 (10.7)
  3 months: 4000 Hz: number analyzed (Participants) | 49
  3 months: 4000 Hz | -26.8 (10.6)
  3 months: 6000 Hz: number analyzed (Participants) | 47
  3 months: 6000 Hz | -31.7 (11.2)
  3 months: 8000 Hz: number analyzed (Participants) | 37
  3 months: 8000 Hz | -30.9 (13.8)
  6 months: 250 Hz: number analyzed (Participants) | 49
  6 months: 250 Hz | -11.9 (11.9)
  6 months: 500 Hz: number analyzed (Participants) | 49
  6 months: 500 Hz | -26.2 (11.3)
  6 months: 750 Hz: number analyzed (Participants) | 43
  6 months: 750 Hz | -30.4 (12.0)
  6 months: 1000 Hz: number analyzed (Participants) | 49
  6 months: 1000 Hz | -28.9 (11.1)
  6 months: 1500 Hz: number analyzed (Participants) | 43
  6 months: 1500 Hz | -28.0 (12.1)
  6 months: 2000 Hz: number analyzed (Participants) | 49
  6 months: 2000 Hz | -26.1 (10.9)
  6 months: 3000 Hz: number analyzed (Participants) | 49
  6 months: 3000 Hz | -27.6 (10.8)
  6 months: 4000 Hz: number analyzed (Participants) | 49
  6 months: 4000 Hz | -30.2 (11.2)
  6 months: 6000 Hz: number analyzed (Participants) | 47
  6 months: 6000 Hz | -31.6 (10.6)
  6 months: 8000 Hz: number analyzed (Participants) | 38
  6 months: 8000 Hz | -33.7 (12.3)
  12 months: 250 Hz: number analyzed (Participants) | 46
  12 months: 250 Hz | -14.7 (12.8)
  12 months: 500 Hz: number analyzed (Participants) | 46
  12 months: 500 Hz | -27.8 (10.9)
  12 months: 750 Hz: number analyzed (Participants) | 40
  12 months: 750 Hz | -31.8 (11.6)
  12 months: 1000 Hz: number analyzed (Participants) | 46
  12 months: 1000 Hz | -31.8 (10.6)
  12 months: 1500 Hz: number analyzed (Participants) | 40
  12 months: 1500 Hz | -31.2 (12.1)
  12 months: 2000 Hz: number analyzed (Participants) | 46
  12 months: 2000 Hz | -28.8 (11.1)
  12 months: 3000 Hz: number analyzed (Participants) | 46
  12 months: 3000 Hz | -29.6 (12.0)
  12 months: 4000 Hz: number analyzed (Participants) | 46
  12 months: 4000 Hz | -33.0 (12.2)
  12 months: 6000 Hz: number analyzed (Participants) | 45
  12 months: 6000 Hz | -35.9 (11.6)
  12 months: 8000 Hz: number analyzed (Participants) | 35
  12 months: 8000 Hz | -38.8 (12.0)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Threshold audiometry 250Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 500Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 750Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1500Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 2000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 3000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 4000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 6000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 8000Hz at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 250Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 12: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 500Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 13: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 750Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 14: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 15: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1500Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 16: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 2000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 17: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 3000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 18: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 4000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 19: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 6000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 20: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 8000Hz at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 21: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 250Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 22: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 500Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 23: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 750Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 24: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 25: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1500Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 26: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 2000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 27: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 3000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 28: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 4000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 29: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 6000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 30: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 8000Hz at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 31: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 250Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 32: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 500Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 33: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 750Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 34: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 35: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 1500Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 36: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 2000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 37: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 3000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 38: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 4000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 39: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 6000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 40: Comparison: Bone-conduction Hearing Device; Threshold audiometry at 8000Hz at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

5. Secondary Outcome: Speech in Quiet at 50, 65 and 80 dB SPL, Unaided Versus OSIA System at 4 Weeks, 3, 6 and 12 Months
Description: The change of hearing performance from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 4 weeks, 3, 6 and 12 months, measured as free-field hearing test Speech in quiet at 50, 65 and 80 dB SPL [% correctly perceived words at 50, 65 and 80 dB SPL] is presented. The change in percent points is presented. A positive value indicates an improved ability to perceive words in quiet at the specified decibel (dB) level a negative value represent an impairment.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months after surgery.
Population: Some of the subjects did not perform the test at one or more visits.
Measure: Mean (Standard Deviation); unit: Percentage of correctly perceived words
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 49
Percentage of correctly perceived words
  4 weeks; 50 dB | 38.0 (27.0)
  4 weeks; 65 dB | 59.8 (28.8)
  4 weeks; 80 dB | 29.3 (30.8)
  3 months: 50 dB | 40.1 (26.8)
  3 months: 65 dB | 60.6 (26.8)
  3 months: 80 dB | 31.8 (31.9)
  6 months: 50 dB: number analyzed (Participants) | 48
  6 months: 50 dB | 46.5 (29.5)
  6 months: 65 dB: number analyzed (Participants) | 48
  6 months: 65 dB | 61.5 (27.7)
  6 months: 80 dB: number analyzed (Participants) | 48
  6 months: 80 dB | 30.7 (33.3)
  12 months: 50 dB: number analyzed (Participants) | 46
  12 months: 50 dB | 57.8 (24.9)
  12 months: 65 dB: number analyzed (Participants) | 46
  12 months: 65 dB | 68.3 (23.6)
  12 months: 80 dB: number analyzed (Participants) | 46
  12 months: 80 dB | 32.7 (32.4)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

6. Secondary Outcome: Adaptive Speech Recognition in Noise, Unaided Versus OSIA System at 4 Weeks, 6 and 12 Months
Description: The change of hearing performance from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 3 months measured as free field hearing test Adaptive speech recognition in noise, is presented. Adaptive speech recognition in noise was measured as Signal to Noise Ratio (SNR). The noise was kept constant at 65 dB SPL and the speech was adapted in dB steps to establish the Speech-to-Noise Ratio (SNR) providing a 50% level of understanding. A ratio of 0 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A negative SNR-value reflects the ability to correctly hear sentences below 65 dB, for example if 50% of the speech is received correctly at 55 dB the SNR value is -10. A positive SNR-value (Speech to Noise Ratio) reflects the ability to correctly hear sentences presented above 65 dB. A lower or more negative score is more desirable and reflects a better hearing in a noisy environment.
Time Frame: Baseline before surgery, 4 weeks, 6 and 12 months after surgery
Population: Some subjects did not perform the test at one or more visits.
Measure: Mean (Standard Deviation); unit: SNR (Speech in Noise Ratio)
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 49
SNR (Speech in Noise Ratio)
  4 weeks | -12.1 (8.1)
  6 months: number analyzed (Participants) | 48
  6 months | -13.7 (8.1)
  12 months: number analyzed (Participants) | 45
  12 months | -13.6 (8.8)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Adaptive speech recognition in noise at 4 weeks with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Adaptive speech recognition in noise at 6 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Adaptive speech recognition in noise at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

7. Secondary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB) at 3 and 12 Months
Description: The change of Ease of communication, Reverberation, Background noise, Aversiveness and a Global score from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 3 and 12 months is presented. All subscales range from 0-100%, total score is the average of all subscales 0-100%, where 0% indicates no problem and 100% indicates always problem. The difference between the unaided and the aided situation is presented. In an ultimate case the unaided value could be 100 and the aided 0, the result is then 100. A positive value indicates an improvement, a negative value an impairment.
Time Frame: Baseline before surgery, 3 and 12 months after surgery
Population: Some of the subjects did not answer some of the questions at one or more visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 48
units on a scale
  3 months: Ease of communication: number analyzed (Participants) | 46
  3 months: Ease of communication | 24.1 (21.7)
  3 months: Background noise: number analyzed (Participants) | 47
  3 months: Background noise | 29.4 (20.0)
  3 months: Reverberation: number analyzed (Participants) | 47
  3 months: Reverberation | 25.8 (23.1)
  3 months: Aversiveness: number analyzed (Participants) | 46
  3 months: Aversiveness | -2.2 (22.3)
  3 months: Global: number analyzed (Participants) | 47
  3 months: Global | 26.1 (18.5)
  12 months: Ease of communication | 24.0 (19.1)
  12 months: Background noise | 29.6 (20.9)
  12 months: Reverberation | 25.4 (25.8)
  12 months: Aversiveness | -3.58 (24.6)
  12 months: Global | 26.3 (18.5)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; APHAB, Ease of communication, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; APHAB, Background noise, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; APHAB, Reverberation, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; APHAB, Aversiveness, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.51, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; APHAB, Global score, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; APHAB, Ease of communication, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; APHAB, Background noise, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; APHAB, Reverberation, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; APHAB, Aversiveness, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.32, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; APHAB, Global score, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

8. Secondary Outcome: Health Utility Index (HUI) at 3 and 12 Months
Description: The change of health status and health related quality of life from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 3 and 12 months using the generic quality of life scale Health Utilities Index (HUI3) is presented. All subscales (comprehensive health state, vision, hearing, speech, ambulation, dexterity, emotion, pain, cognition) range from 0-1. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. The difference between the unaided and the aided situation is presented. In an ultimate case the unaided value could be 0 and the aided 1, the result is then 1.0. A positive value indicates an improved quality of life, a negative value indicates impaired quality of life.
Time Frame: Baseline before surgery and 3 and 12 months after surgery
Population: Some of the subjects did not answer all questions in the questionnaire at one or both time-points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 48
units on a scale
  3 months: comprehensive health state: number analyzed (Participants) | 42
  3 months: comprehensive health state | 0.081 (0.227)
  3 months: Vision: number analyzed (Participants) | 46
  3 months: Vision | -0.006 (0.035)
  3 months: Hearing: number analyzed (Participants) | 44
  3 months: Hearing | 0.173 (0.324)
  3 months: Speech | 0.033 (0.129)
  3 months: Ambulation | -0.018 (0.063)
  3 months: Dexterity | 0.000 (0.000)
  3 months: Emotion | 0.016 (0.120)
  3 months: Cognition | 0.013 (0.088)
  3 months: Pain | 0.007 (0.258)
  12 months: comprehensive health state: number analyzed (Participants) | 42
  12 months: comprehensive health state | 0.058 (0.243)
  12 months: Vision: number analyzed (Participants) | 47
  12 months: Vision | -0.011 (0.055)
  12 months: Hearing: number analyzed (Participants) | 42
  12 months: Hearing | 0.149 (0.300)
  12 months: Speech | 0.062 (0.136)
  12 months: Ambulation | -0.024 (0.094)
  12 months: Dexterity | -0.011 (0.122)
  12 months: Emotion | 0.004 (0.144)
  12 months: Cognition: number analyzed (Participants) | 47
  12 months: Cognition | 0.001 (0.125)
  12 months: Pain | -0.029 (0.334)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; HUI Comprehensive health state at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.026, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; HUI Vision attribute at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.50, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; HUI Hearing attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.0008, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; HUI Speech attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.082, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; HUI Ambulation attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.13, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; HUI Dexterity attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.9, Wilcoxon Signed Rank test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; HUI Emotion attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.43, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; HUI Cognition attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.31, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; HUI Pain attribute, at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.72, Wilcoxon Signed Rank test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; HUI Comprehensive Health State attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.13, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Bone-conduction Hearing Device; HUI Vision attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.23, Wilcoxon Signed Rank test
Statistical Analysis 12: Comparison: Bone-conduction Hearing Device; HUI Hearing attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.0026, Fisher's non-parametric permutation test
Statistical Analysis 13: Comparison: Bone-conduction Hearing Device; HUI Speech attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.0024, Fisher's non-parametric permutation test
Statistical Analysis 14: Comparison: Bone-conduction Hearing Device; HUI Ambulation attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.16, Fisher's non-parametric permutation test
Statistical Analysis 15: Comparison: Bone-conduction Hearing Device; HUI Dexterity attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.16, Fisher's non-parametric permutation test
Statistical Analysis 16: Comparison: Bone-conduction Hearing Device; HUI Emotion attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.85, Fisher's non-parametric permutation test
Statistical Analysis 17: Comparison: Bone-conduction Hearing Device; HUI Cognition attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 1.0, Fisher's non-parametric permutation test
Statistical Analysis 18: Comparison: Bone-conduction Hearing Device; HUI Pain attribute, at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p = 0.56, Fisher's non-parametric permutation test

9. Secondary Outcome: Speech, Spatial and Qualities of Hearing Scale (SSQ) at 3 and 12 Months
Description: The change of speech, spatial and hearing experiences from the unaided hearing situation before surgery to the aided hearing situation with the OSIA System at 3 and 12 months using the SSQ scale is presented. All subscales (speech, spatial, quality) range from 0 to 10, where 0 represents "can not hear at all", and 10 "hear perfectly". Total score is a average of the subscales. A positive value indicates improved hearing, a negative value indicates impaired hearing.
Time Frame: Baseline before surgery and 3 and 12 months after surgery
Population: Some of the subjects did not answer all questions at one or both visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 48
units on a scale
  3 months: Total score: number analyzed (Participants) | 47
  3 months: Total score | 2.57 (2.01)
  3 months: Speech score: number analyzed (Participants) | 47
  3 months: Speech score | 2.91 (2.19)
  3 months: Spatial score: number analyzed (Participants) | 47
  3 months: Spatial score | 2.85 (2.50)
  3 months: Quality score | 1.88 (2.38)
  12 months: Total score: number analyzed (Participants) | 47
  12 months: Total score | 2.69 (1.75)
  12 months: Speech score: number analyzed (Participants) | 47
  12 months: Speech score | 2.94 (1.94)
  12 months: Spatial score: number analyzed (Participants) | 47
  12 months: Spatial score | 2.95 (2.52)
  12 months: Quality score | 2.13 (2.30)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; SSQ Total score at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; SSQ Speech score at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; SSQ Spatial score at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; SSQ Quality score at 3 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; SSQ Total score at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; SSQ Speech score at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; SSQ Spatial score at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; SSQ Quality score at 12 months with the Osia system vs Unaided at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

10. Secondary Outcome: Hearing Performance: Threshold Audiometry PTA4, With Reference Device BP110
Description: The change of hearing performance with the OSIA System at 4 weeks, 3, 6 and 12 months compared to the pre-operative aided situation with BP110 on softband, measured as free-field hearing test; Threshold audiometry PTA4 (mean of 500, 1000, 2000 and 4000 Hz) is presented. The units reported for PTA4 are decibels (dB). A lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months.
Population: Some of the subjects did not perform a PTA4 measurement at one or more visits.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
dB
  4 weeks | -3.16 (5.68)
  3 months: number analyzed (Participants) | 49
  3 months | -3.82 (5.94)
  6 months: number analyzed (Participants) | 49
  6 months | -5.72 (5.84)
  12 months: number analyzed (Participants) | 46
  12 months | -7.85 (6.35)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry PTA4 with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry PTA4 with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry PTA4 with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry PTA4 with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

11. Secondary Outcome: Hearing Performance: Threshold Audiometry Individual Frequences With Reference Device BP110
Description: The change of hearing performance with the OSIA System at 4 weeks, 3, 6 and 12 months compared to the pre-operative aided situation with BP110 on softband, measured as free-field hearing test; Threshold audiometry individual frequencies (0.25, 0.5, 0.75, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0 and 8.0 kHz) is presented. The units reported are decibels (dB). A lower or more negative score is more desirable and reflects a better ability to hear softer sounds.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months after surgery.
Population: Some of the subjects did not perform all measurements at all visits.
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
dB
  4 weeks: 250 hz | 3.58 (10.98)
  4 weeks: 500 Hz | -2.22 (9.15)
  4 weeks: 750 Hz: number analyzed (Participants) | 43
  4 weeks: 750 Hz | -3.30 (8.49)
  4 weeks: 1000 Hz | 0.42 (6.65)
  4 weeks: 1500 Hz: number analyzed (Participants) | 44
  4 weeks: 1500 Hz | -0.48 (8.39)
  4 weeks: 2000 Hz | -2.62 (7.66)
  4 weeks: 3000 Hz | -3.18 (7.86)
  4 weeks: 4000 Hz | -8.20 (9.58)
  4 weeks: 6000 Hz | -12.5 (10.3)
  4 weeks: 8000 Hz: number analyzed (Participants) | 41
  4 weeks: 8000 Hz | -16.4 (17.3)
  3 months: 250 Hz: number analyzed (Participants) | 49
  3 months: 250 Hz | 3.20 (9.19)
  3 months: 500 Hz: number analyzed (Participants) | 49
  3 months: 500 Hz | -2.69 (8.86)
  3 months: 750 Hz: number analyzed (Participants) | 43
  3 months: 750 Hz | -2.86 (8.66)
  3 months: 1000 Hz: number analyzed (Participants) | 49
  3 months: 1000 Hz | -0.47 (7.22)
  3 months: 1500 Hz: number analyzed (Participants) | 43
  3 months: 1500 Hz | -1.19 (7.82)
  3 months: 2000 Hz: number analyzed (Participants) | 49
  3 months: 2000 Hz | -3.37 (8.15)
  3 months: 3000 Hz: number analyzed (Participants) | 49
  3 months: 3000 Hz | -4.57 (9.11)
  3 months: 4000 Hz: number analyzed (Participants) | 49
  3 months: 4000 Hz | -8.73 (10.07)
  3 months: 6000 Hz: number analyzed (Participants) | 48
  3 months: 6000 Hz | -15.0 (9.9)
  3 months: 8000 Hz: number analyzed (Participants) | 40
  3 months: 8000 Hz | -18.1 (18.4)
  6 months: 250 Hz: number analyzed (Participants) | 49
  6 months: 250 Hz | 2.10 (8.70)
  6 months: 500 Hz: number analyzed (Participants) | 49
  6 months: 500 Hz | -4.69 (8.90)
  6 months: 750 Hz: number analyzed (Participants) | 43
  6 months: 750 Hz | -4.70 (7.90)
  6 months: 1000 Hz: number analyzed (Participants) | 49
  6 months: 1000 Hz | -1.67 (7.03)
  6 months: 1500 Hz: number analyzed (Participants) | 43
  6 months: 1500 Hz | -4.00 (7.23)
  6 months: 2000 Hz: number analyzed (Participants) | 49
  6 months: 2000 Hz | -4.61 (8.29)
  6 months: 3000 Hz: number analyzed (Participants) | 49
  6 months: 3000 Hz | -5.76 (8.06)
  6 months: 4000 Hz: number analyzed (Participants) | 49
  6 months: 4000 Hz | -11.9 (10.4)
  6 months: 6000 Hz: number analyzed (Participants) | 48
  6 months: 6000 Hz | -14.4 (10.7)
  6 months: 8000 Hz: number analyzed (Participants) | 41
  6 months: 8000 Hz | -20.7 (17.6)
  12 months: 250 Hz: number analyzed (Participants) | 46
  12 months: 250 Hz | -0.39 (9.81)
  12 months: 500 Hz: number analyzed (Participants) | 46
  12 months: 500 Hz | -5.91 (8.79)
  12 months: 750 Hz: number analyzed (Participants) | 40
  12 months: 750 Hz | -5.75 (8.65)
  12 months: 1000 Hz: number analyzed (Participants) | 46
  12 months: 1000 Hz | -4.07 (7.98)
  12 months: 1500 Hz: number analyzed (Participants) | 40
  12 months: 1500 Hz | -6.73 (8.21)
  12 months: 2000 Hz: number analyzed (Participants) | 46
  12 months: 2000 Hz | -6.80 (8.33)
  12 months: 3000 Hz: number analyzed (Participants) | 46
  12 months: 3000 Hz | -7.61 (9.13)
  12 months: 4000 Hz: number analyzed (Participants) | 46
  12 months: 4000 Hz | -14.6 (10.8)
  12 months: 6000 Hz: number analyzed (Participants) | 46
  12 months: 6000 Hz | -18.6 (11.4)
  12 months: 8000 Hz: number analyzed (Participants) | 38
  12 months: 8000 Hz | -26.5 (17.3)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 250Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.025, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 500Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.096, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 750Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.015, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.67, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1500Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.73, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 2000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.019, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 3000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0046, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 4000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 6000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 8000Hz with Osia at 4 week vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 250Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.019, Fisher's non-parametric permutation test
Statistical Analysis 12: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 500Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.040, Fisher's non-parametric permutation test
Statistical Analysis 13: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 750Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.037, Fisher's non-parametric permutation test
Statistical Analysis 14: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.67, Fisher's non-parametric permutation test
Statistical Analysis 15: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1500Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.34, Fisher's non-parametric permutation test
Statistical Analysis 16: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 2000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0048, Fisher's non-parametric permutation test
Statistical Analysis 17: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 3000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0008, Fisher's non-parametric permutation test
Statistical Analysis 18: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 4000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 19: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 6000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 8000Hz with Osia at 3 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 21: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 250Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.10, Fisher's non-parametric permutation test
Statistical Analysis 22: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 500Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0007, Fisher's non-parametric permutation test
Statistical Analysis 23: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 750Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0003, Fisher's non-parametric permutation test
Statistical Analysis 24: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.11, Fisher's non-parametric permutation test
Statistical Analysis 25: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1500Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 26: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 2000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 27: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 3000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 28: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 4000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 29: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 6000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 30: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 8000Hz with Osia at 6 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 31: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 250Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.80, Fisher's non-parametric permutation test
Statistical Analysis 32: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 500Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 33: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 750Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 34: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p = 0.0010, Fisher's non-parametric permutation test
Statistical Analysis 35: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 1500Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 36: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 2000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 37: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 3000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 38: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 4000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 39: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 6000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 40: Comparison: Bone-conduction Hearing Device; Hearing performance: threshold audiometry 8000Hz with Osia at 12 months vs the reference device BP110 on a softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

12. Secondary Outcome: Speech in Quiet at 50, 65 and 80 dB SPL, With Reference Device BP110
Description: The change of hearing performance with the OSIA System at 4 weeks, 3, 6 and 12 months compared to the pre-operative aided situation with BP110 on softband measured as free-field hearing test; Speech in quiet [% correctly perceived words at 50, 65 and 80 dB SPL]. The change in percent points is presented. A positive value indicates an improved ability to perceive words in quiet at the specified decibel (dB) level a negative value represent an impairment.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months after surgery.
Population: Some of the subjects did not perform all measurements at all visits.
Measure: Mean (Standard Deviation); unit: Percentage of correctly perceived words
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 48
Percentage of correctly perceived words
  4 weeks: 50 dB SPL | 2.40 (24.81)
  4 weeks: 65 dB SPL | 6.65 (19.58)
  4 weeks: 80 dB SPL | 1.17 (7.34)
  3 months: 50 dB SPL | 5.17 (26.16)
  3 months: 65 dB SPL | 7.48 (21.39)
  3 months: 80 dB SPL | 1.77 (8.35)
  6 months: 50 dB SPL | 10.3 (24.4)
  6 months: 65 dB SPL | 7.73 (22.56)
  6 months: 80 dB SPL | 0.875 (10.02)
  12 months: 50 dB SPL: number analyzed (Participants) | 46
  12 months: 50 dB SPL | 20.7 (29.5)
  12 months: 65 dB SPL: number analyzed (Participants) | 46
  12 months: 65 dB SPL | 13.9 (22.3)
  12 months: 80 dB SPL: number analyzed (Participants) | 46
  12 months: 80 dB SPL | 3.61 (10.45)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB SPL with Osia at 4 weeks vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.51, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB SPL with Osia at 4 weeks vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.021, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB SPL with Osia at 4 weeks vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.29, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB SPL with Osia at 3 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.18, Fisher's non-parametric permutation test
Statistical Analysis 5: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB SPL with Osia at 3 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.017, Fisher's non-parametric permutation test
Statistical Analysis 6: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB SPL with Osia at 3 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.16, Fisher's non-parametric permutation test
Statistical Analysis 7: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB SPL with Osia at 6 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.0051, Fisher's non-parametric permutation test
Statistical Analysis 8: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB SPL with Osia at 6 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.021, Fisher's non-parametric permutation test
Statistical Analysis 9: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB SPL with Osia at 6 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.56, Fisher's non-parametric permutation test
Statistical Analysis 10: Comparison: Bone-conduction Hearing Device; Speech in quiet at 50dB SPL with Osia at 12 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 11: Comparison: Bone-conduction Hearing Device; Speech in quiet at 65dB SPL with Osia at 12 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 12: Comparison: Bone-conduction Hearing Device; Speech in quiet at 80dB SPL with Osia at 12 months vs reference device BP110 on softband att visit 1; Test type: Superiority; p = 0.041, Wilcoxon Signed Rank test

13. Secondary Outcome: Adaptive Speech Recognition in Noise, With Reference Device BP110
Description: The change of hearing performance with the OSIA System at 4 weeks, 3, 6 and 12 months compared to the pre-operative aided situation with BP110 on softband;measured with free field hearing test Adaptive speech recognition in noise which was measured as signal to noise ratio (SNR). The noise was kept constant at 65 dB SPL and the speech was adapted in dB steps to establish the speech-to-noise ratio (SNR) providing a 50% level of understanding. A ratio of 0 reflects the ability to correctly hear sentences at 65 dB, in the presence of 65 dB background noise. A negative SNR-value reflects the ability to correctly hear sentences below 65 dB. A positive SNR-value reflects the ability to correctly hear sentences presented above 65 dB. A lower or more negative score is more desirable and represent a better hearing in a noisy environment.
Time Frame: Baseline before surgery, 4 weeks, 3, 6 and 12 months after surgery.
Population: Some of the subjects did not perform the test at all visits.
Measure: Mean (Standard Deviation); unit: SNR
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 47
SNR
  4 weeks | -6.12 (6.92)
  3 months | -7.19 (6.80)
  6 months: number analyzed (Participants) | 46
  6 months | -7.91 (6.80)
  12 months: number analyzed (Participants) | 44
  12 months | -7.54 (7.99)
Statistical Analysis 1: Comparison: Bone-conduction Hearing Device; Adaptive Speech Recognition in Noise with Osia at 4 weeks vs reference device BP110 on softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 2: Comparison: Bone-conduction Hearing Device; Adaptive Speech Recognition in Noise with Osia at 3 months vs reference device BP110 on softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 3: Comparison: Bone-conduction Hearing Device; Adaptive Speech Recognition in Noise with Osia at 6 months vs reference device BP110 on softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test
Statistical Analysis 4: Comparison: Bone-conduction Hearing Device; Adaptive Speech Recognition in Noise with Osia at 12 months vs reference device BP110 on softband at visit 1; Test type: Superiority; p < 0.0001, Fisher's non-parametric permutation test

14. Secondary Outcome: Surgical Information: Time of Surgery
Description: Surgery time in minutes between first incision and last suture
Time Frame: Visit 2, surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
minutes | 97.2 (27.8)

15. Secondary Outcome: Soft Tissue Thickness
Description: Surgical information: Soft tissue thickness was measured in mm
Time Frame: Visit 2, surgery
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
mm | 6.00 (1.30)

16. Secondary Outcome: Soft Tissue Reduction
Description: Surgical information: a question was asked if soft tissue reduction had been performed. Could be answered by ticking a box for "Yes" or "No".
Time Frame: Visit 2, surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
Participants
  Yes | 10
  No | 41

17. Secondary Outcome: Bone Polishing/Removal at Implant Site
Description: Surgical information: a question is asked if bone polishing/removal at Implant site has been performed. Yes or No can be ticked.
Time Frame: Visit 2, surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
Participants
  Yes | 42
  No | 9

18. Secondary Outcome: Type of Anaesthesia
Description: Surgical information: a question is asked which type of anaesthesia has been used: local or general can be ticked.
Time Frame: Visit 2, surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
Participants
  General | 51
  Local | 0

19. Secondary Outcome: Location of BI300 Implant
Description: Surgical information: where is the location of the BI300 implant, measured in two different ways:
  Alternative 1 used for the first 6 subjects: Location from the ear channel in mm.
  Alternative 2 used for the rest of the population 45 subjects, after an amendment: measured in mm horizontally and vertically from ear channel. and the distance in mm between the receiver and the coil.
  Value 9.64 mm vertically from ear channel is correct.
Time Frame: Visit 2, surgery
Population: Localization of the BI300 implant measured in two different ways; 6 subjects with alternative 1, 45 subjects with alternative 2.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
mm
  Alt 1: distance from the ear channel: number analyzed (Participants) | 6
  Alt 1: distance from the ear channel | 48.3 (10.3)
  9.64Alt 2: horizontally from ear channel: number analyzed (Participants) | 45
  9.64Alt 2: horizontally from ear channel | 40.0 (17.9)
  Alt 2: vertically from the ear channel: number analyzed (Participants) | 45
  Alt 2: vertically from the ear channel | 9.64 (9.20)
  Alt 2: distance between receiver and coil: number analyzed (Participants) | 45
  Alt 2: distance between receiver and coil | 54.4 (13.8)

20. Secondary Outcome: Incision Type
Description: Surgical information: a question was asked regarding what type of incision had been used; C-shaped flap, posterior based flap or other could be ticked.
Time Frame: Visit 2, surgery
Population: For two subjects two alternatives were checked.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 51
Participants
  C-shaped flap | 30
  Poesterior flap | 1
  Other | 22

21. Secondary Outcome: Daily Usage Time of Sound Processor
Description: Sound processor usage time measured as hours per day.
Time Frame: 6 weeks, 3, 6 and 12 months
Population: Some of the subjects did not answer the question at all visits.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
hours per day
  6 weeks: number analyzed (Participants) | 48
  6 weeks | 10.7 (3.8)
  3 months: number analyzed (Participants) | 47
  3 months | 10.5 (4.3)
  6 months | 10.6 (4.6)
  12 months: number analyzed (Participants) | 47
  12 months | 11.3 (3.6)

22. Secondary Outcome: Comfort
Description: Comfort of sound processor measured with a visual analogue scale where 0% is defined as no comfort at all and 100% as most comfortable imaginable, i.e. minimum 0, maximum 100.
Time Frame: 6 weeks, 3, 6 and 12 months
Population: Some of the subjects did not answer the question at all visits.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
units on a scale
  6 weeks: number analyzed (Participants) | 49
  6 weeks | 77.3 (18.6)
  3 months: number analyzed (Participants) | 46
  3 months | 80.8 (16.6)
  6 months: number analyzed (Participants) | 48
  6 months | 78.2 (20.1)
  12 months: number analyzed (Participants) | 47
  12 months | 80.9 (16.2)

23. Secondary Outcome: Magnet Choice
Description: Available magnet strengths: 1/2, 1, 2, 3, 4, 5 or 6, where 1/2 is the weakest and 6 the strongest.
Time Frame: 4, 6 weeks, 3, 6 and 12 months
Population: Some of the subjects did not perform all visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
Participants
  4 weeks: strength 1/2 | 0
  4 weeks: strength 1 | 1
  4 weeks: strength 2 | 11
  4 weeks: strength 3 | 13
  4 weeks: strength 4 | 12
  4 weeks: strength 5 | 8
  4 weeks: strength 6 | 5
  6 weeks strength 1/2: number analyzed (Participants) | 49
  6 weeks strength 1/2 | 0
  6 weeks strength 1: number analyzed (Participants) | 49
  6 weeks strength 1 | 1
  6 weeks strength 2: number analyzed (Participants) | 49
  6 weeks strength 2 | 10
  6 weeks strength 3: number analyzed (Participants) | 49
  6 weeks strength 3 | 11
  6 weeks strength 4: number analyzed (Participants) | 49
  6 weeks strength 4 | 13
  6 weeks strength 5: number analyzed (Participants) | 49
  6 weeks strength 5 | 9
  6 weeks strength 6: number analyzed (Participants) | 49
  6 weeks strength 6 | 5
  3 months strength 1/2 | 0
  3 months strength 1 | 1
  3 months strength 2 | 12
  3 months strength 3 | 10
  3 months strength 4 | 14
  3 months strength 5 | 8
  3 months strength 6 | 5
  6 months strength 1/2 | 0
  6 months strength 1 | 2
  6 months strength 2 | 11
  6 months strength 3 | 11
  6 months strength 4 | 13
  6 months strength 5 | 10
  6 months strength 6 | 3
  12 months strength 1/2: number analyzed (Participants) | 48
  12 months strength 1/2 | 0
  12 months strength 1: number analyzed (Participants) | 48
  12 months strength 1 | 2
  12 months strength 2: number analyzed (Participants) | 48
  12 months strength 2 | 12
  12 months strength 3: number analyzed (Participants) | 48
  12 months strength 3 | 10
  12 months strength 4: number analyzed (Participants) | 48
  12 months strength 4 | 11
  12 months strength 5: number analyzed (Participants) | 48
  12 months strength 5 | 10
  12 months strength 6: number analyzed (Participants) | 48
  12 months strength 6 | 3

24. Secondary Outcome: Softpad Use
Description: A question was asked if the subjects used softpads; yes or no could be ticked.
Time Frame: 6 weeks, 3, 6 and 12 months
Population: Some of the subjects did not answer the question at all visits.
Measure: Count of Participants; unit: Participants
Arm/Group | Bone-conduction Hearing Device
Number analyzed (Participants) | 50
Participants
  6 weeks: yes: number analyzed (Participants) | 48
  6 weeks: yes | 1
  6 weeks: no: number analyzed (Participants) | 48
  6 weeks: no | 47
  3 months: yes: number analyzed (Participants) | 49
  3 months: yes | 4
  3 months: no: number analyzed (Participants) | 49
  3 months: no | 45
  6 months: yes | 0
  6 months: no | 50
  12 months: yes: number analyzed (Participants) | 47
  12 months: yes | 3
  12 months: no: number analyzed (Participants) | 47
  12 months: no | 44

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bone-conduction Hearing Device
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 2/51
Other Adverse Events (participants affected / at risk) | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone-conduction Hearing Device (N=51)
Wound infection (Infections and infestations) | 1 (51) — Infection at implant site starting shortly after surgery, lead to explantation.
Infection and infestations (Infections and infestations) | 1 (51) — One subject was hospitalized three days due to an influenza infection.
Atrial fibrilation (Cardiac disorders) | 1 (51) — 0ne subject was treated for persistent atrial fibrillation.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bone-conduction Hearing Device (N=51)
Hearing impaired (Ear and labyrinth disorders) | 18 (19)
General disorders and administration site conditions other (General disorders) | 14 (15)
Otitis externa (Infections and infestations) | 4 (4)
Headache (Nervous system disorders) | 3 (3)
Nervous system disorders other (Nervous system disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/35/NCT03086135/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-16): https://cdn.clinicaltrials.gov/large-docs/35/NCT03086135/SAP_001.pdf